CLINICAL TRIAL: NCT06857994
Title: The Association Between Cognitive Function and Diabetic Neuropathy in Individuals With Type 2 Diabetes
Brief Title: The Association Between Cognitive Function and Neuropathy in Individuals With Type 2 Diabetes
Acronym: ASCEND
Status: Recruiting | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: H-24014649
Record Dates: First submitted 2025-01-22; First posted 2025-03-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Diabetic Neuropathy; Cardiovascular Autonomic Neuropathy; Cognitive Impairment; Diabetes Type 2
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples with DNA: Blood samples (serum, plasma, buffy coat are frozen) Samples without DNA: Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 2 Diabetes and No Neuropathy: This group consists of individuals who meet the inclusion and exclusion criteria and have normal peripheral and cardiovascular autonomic nerve function.
- Type 2 Diabetes with Peripheral Neuropathy: This group consists of individuals who meet the inclusion and exclusion criteria and have peripheral neuropathy and normal cardiovascular autonomic nerve function.
- Type 2 Diabetes with Cardiovascular Autonomic Neuropathy: This group consists of individuals who meet the inclusion and exclusion criteria and have cardiovascular autonomic neuropathy. They can have a normal or abnormal peripheral nerve test.
- Controls (No Type 2 Diabetes): This group consists of individuals who meet the inclusion and exclusion criteria for controls.

SUMMARY:
The goal of this observational study is to evaluate whether individuals with different types of diabetic neuropathy (peripheral and cardiovascular autonomic neuropathy) are at an increased risk of cognitive impairment and to investigate the potential reasons for this association.

The primary research question is: Is diabetic peripheral and cariovascular autonomic neuropathy in type 2 diabetes associated with cognitive decline?

To address this question, the study will include individuals with and without type 2 diabetes. All participants will undergo comprehensive neuropathy assessments, neuropsychological evaluations and blood biomarker analysis. In addition, some individuals will undergo structural and functional brain MRI.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a chronic disease with complications that affect various organs over time. While certain complications have been well- established for decades, recent research points to the brain as an important site of diabetes-associated damage. This aligns with the growing awareness of the cognitive impact of diabetes. Diabetes is associated with mild to moderate alterations in cognitive functions across diverse age groups and an increased risk of developing dementia. The precise mechanism underlying these associations remains elusive, but some studies suggest that impaired peripheral nerve function correlates with negative cognitive outcomes and may be associated with structural and functional brain changes. Since diabetic neuropathy is one of the most common complications of diabetes, it might contribute to an increased dementia risk.

ASCEND is a clinical descriptive study that aims to evaluate the association between diabetic neuropathy and cognitive function in individuals with type 2 diabetes (compared to controls without diabetes). The study comprises the following visits:

* Screening visit
* Neuropathy assessment and neuropsychological testing visit
* Structural and functional MRI (only a subset of participants)

The neuropathy assessment will include the following measures:

* Peripheral vibration sensation (biothesiometer)
* Cardiovascular autonomic neuropathy (Vagus device) both resting heart rate variability and cardiovascular reflex tests
* Nerve conduction velocity and amplitude of the Sural nerves by DPN-check
* Light touch and pain sensation (10 g monofilament and 40g needle)
* Peripheral small-fiber sympathetic function (Sudoscan device)
* Cold and warm sensation of foot and lower leg

The neuropsychological test will include the following:

* Rey Auditory Verbal Learning Test (RAVLT)
* Trail Making Test (TMT) part A and B
* Symbol Digit Modalities Test (SDMT)
* RBANS Digit Span forward (Version A)
* Wechsler Adult Intelligence Scale III Letter-Number Sequencing test (WAIS-LNS)
* Verbal Fluency test (letters S and D)
* Grooved Pegboard
* Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automated Battery (CANTAB) using A' (RVP-A) and mean latency for correct responses

ELIGIBILITY:
Since the study includes both individuals with and without diabetes, there are two sets of inclusion criteria. Exclusion criteria apply to both indivdiuals with and without diabetes.

Inclusion Criteria:

For individuals with type 2 diabetes:

* Age >= 65 years
* Type 2 Diabetes diagnosis (defined according to the criteria from World Health Organization) for more than 5 years
* BMI <= 35
* Stable diabetes treatment for at least 8 weeks (adjustments of already prescribed insulin doses are accepted)
* Plasma hemoglobin ≥ 8.00 mmol/L (male) or ≥ 6.4 mmol/L (female)
* Speaks and understands Danish (required for the cognitive tests)
* Informed and written consent

For individuals without type 2 diabetes:

* Age ≥ 65 years
* Not diagnosed with T2D diagnosis (defined according to criteria from World Health Organization (WHO))
* Speaks and understands Danish (required for the cognitive tests)
* Informed and written consent

Exclusion Criteria (all individuals):

* Any medical condition which, based on investigators assessment, challenges or hinders participation in cognitive screening, impedes compliance with the study protocol or evaluation of results, including but not limited to psychiatric disorders, neurological disorders, chronic pain disorders etc.
* Significant history of alcoholism or drug/chemical substance abuse as per the investigator's judgement.
* Individuals in active laser treatment for retinopathy, atrial fibrillation, atrial flutter, or pacemakers since these cannot take part in CAN measurements.
* Individuals unable to take part in the MRI because of e.g., metallic objects in the body or severe claustrophobia.
* Individuals who do not wish to be informed about accidental findings by MR.
* Diagnosis of dementia (ICD F00-F03) or participants who have previously been referred to a dementia clinic.
* Severe hypoglycemic events during the past 6 months requiring medical assistance.
* Severe renal insufficiency as eGFR ≤ 30 ml/min/1.73 m2
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range of 90-150 mmHg for systolic and 50-100 for diastolic.
* Active or recent (≤ 12 months) malignant disease as judged by the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Cisgender people who identify with the gender that aligns with the sex they were assigned at birth.
Study Population: Individuals with type 2 diabetes will be recruited among the participants in a former study at teno Diabetes Center Copenhagen, Denmark (DANES-study) who at the time of participation accepted to be contacted again regarding other research projects.
  Healthy controls will be recruited among persons who have previously participated in studies at SDCC and at the time of participation accepted to be contacted again regarding other research projects. In addition to this, participants will be sought by physical advertisements in the local area, through Facebook groups (all posts that are part of the campaigns, will be created, so it is not possible to comment or tag on them) and through forskningnu.dk.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive composite score (global score) | Baseline (only measured once)
  The global score is based on the scores the neuropsychological test battery. The tests are grouped based on cognitive domains and the global cognitive score is assessed by the mean of individual component z-scores.
  The neuropsychological test battery will include the following:
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT) part A and B
  * Symbol Digit Modalities Test (SDMT)
  * RBANS Digit Span forward (Version A)
  * Wechsler Adult Intelligence Scale III Letter-Number Sequencing test (WAIS-LNS)
  * Verbal Fluency test (letters S and D)
  * Grooved Pegboard
  * Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automated Battery (CANTAB) using A' (RVP-A) and mean latency for correct responses

SECONDARY OUTCOMES:
Cognitive domain scores | Baseline (only measured once)
  The cognitive domain scores are based on the scores from the neuropsychological test battery. The cognitive domain score is assessed by the mean of individual component z-scores.
  The neuropsychological test battery will include the following:
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT) part A and B
  * Symbol Digit Modalities Test (SDMT)
  * RBANS Digit Span forward (Version A)
  * Wechsler Adult Intelligence Scale III Letter-Number Sequencing test (WAIS-LNS)
  * Verbal Fluency test (letters S and D)
  * Grooved Pegboard
  * Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automated Battery (CANTAB) using A' (RVP-A) and mean latency for correct responses
The reduction in gray matter volume in primary somatosensory cortex (S1), primary motor cortex (M1) and hippocampus | Baseline (only measured once)
  Structural brain MRI
Differences in whiter matter hyperintensities and microbleeds | Baseline (only measured once)
  Structural brain MRI
Differences in resting state BOLD (Blood oxygenation level dependent) signal | Baseline (only measured once)
  Functional brain MRI
Differences in BOLD (Blood oxygenation level dependent) signal during n-back memory task | Baseline (only measured once)
  Functional MRI

OTHER OUTCOMES:
Self-rated health-related quality of life, assessed by Short Form 36 (questionnaire) | Baseline (only measured once)
  Short Form 36 (SF-36) is a health-related questionnarie. The questionnaire consits of eight domains with scores range from 0 to 100. A score of 0 indicates the worst health status, while a score of 100 indicates the best possible health status.
The difference in diabetes distress, assessed by Problem Areas in Diabetes (PAID) 20 | Baseline (only measured once)
  Scores range from 0 - 100, higer scores indicate worse outcome.
The difference in measured levels of blood-based biomarkers of peripheral and central nerve damage | Baseline (only measured once)
  Interleukins (IL-1β, IL-6, IL-8, IL-10), tumor necrosis factor-alpha (TNF-α), interferon-gamma (IFN-γ), amyloid-beta, total tau (t-tau), phosphorylated tau (p-tau), neurofilaments (NfL, NfM, NfH, a-internexin, peripherin), glial fibrillary acidic protein (GFAP), neuronally derived plasma exosomes, matrix metalloproteinases, S100B and glycocalyx markers (keratan sulfate, chondroitin sulfate, heparan sulfate, hyaluronic acid, CD44, syndecan-1-4, glypican-1, BiGlycan).

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No